CLINICAL TRIAL: NCT01020487
Title: A Phase 3, Prospective, Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Pharmacokinetics, Safety and Efficacy of Paricalcitol Capsules in Decreasing Serum Intact Parathyroid Hormone Levels in Pediatric Subjects Ages 10 to 16 Years With Moderate to Severe Chronic Kidney Disease
Brief Title: Safety and Efficacy of Paricalcitol Capsules in Decreasing Serum Parathyroid Hormone Levels in Children Aged 10-16 With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-149; 2010-019439-37 (EudraCT Number)
Record Dates: First submitted 2009-11-13; First posted 2009-11-24 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-02

CONDITIONS: Chronic Kidney Disease Stage 3 and 4
Keywords: Reduction of parathyroid hormone levels in pediatric patients with Chronic Kidney Disease Stage 3 and 4
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Paricalcitol (Experimental): Participants received a single 3 µg dose of paricalcitol capsules on Study Day 1.
  Interventions: Drug: Paricalcitol
- Part 2: Placebo (Placebo Comparator): Participants received placebo capsules three times a week (TIW) for 12 weeks during the double-blind treatment phase. From Weeks 12 to 24 participants received open-label paricalcitol at an initial dose of 1 µg three times a week. Doses could be increased in 1 μg increments every 4 weeks based on chemistry evaluations to target Kidney Disease Outcomes Quality Initiatives (KDOQI) target levels.
  Interventions: Drug: Paricalcitol; Drug: Placebo
- Part 2: Paricalcitol (Experimental): Participants received paricalcitol three times a week for 12 weeks during the double-blind treatment period and during the open-label period (Weeks 12-24). The initial dose of paricalcitol was 1 µg TIW. Doses could be increased in 1 μg increments every 4 weeks based on chemistry evaluations to target KDOQI target levels.
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol capsules taken with water.
  Other Names: Zemplar
Drug: Placebo — Placebo capsules taken with water
  Arms: Part 2: Placebo

SUMMARY:
Part 1: To determine the safety, tolerability, and pharmacokinetics of a single dose of 3 μg paricalcitol capsules in children ages 10 to 16 years with moderate to severe chronic kidney disease (CKD Stages 3 and 4).

Part 2: To determine the safety and efficacy of paricalcitol capsules as compared to placebo in decreasing serum intact parathyroid hormone (iPTH) in children ages 10 to 16 years with moderate to severe chronic kidney disease with an initial 12 weeks of double-blinded study drug followed by a minimum of 12 weeks of open-label active drug.

DETAILED DESCRIPTION:
The study consists of two parts. Part 1 is an open-label single-dose, non-fasting, multicenter study to evaluate the pharmacokinetics (PK) of paricalcitol capsules in 12 children ages 10 to 16 years with CKD Stages 3 and 4. Part 2 of this study will be conducted as a 12 week randomized double-blind, placebo-controlled study, followed by 12 weeks open-label treatment. Participants active or enrolled under amendment 5 will enter a follow-up period and have study visits every 4 weeks until the final participant reaches Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Subject has chronic kidney disease Stage 3 or 4 as determined by estimated glomerular filtration rate (15 to 59 mL/min/1.73 m²) at Screening.
* Subject is not expected to begin dialysis for at least 6 months (in the opinion of the investigator).
* For entry into the Washout Period (for subjects who are currently on a vitamin D receptor activator [VDRA] and need to complete a 2 to 4 week washout), the subject must satisfy the following criteria based on the Screening laboratory values:

  * estimated glomerular filtration rate between 15 to 59 mL/min/1.73 m².
  * iPTH measurement that is greater than or equal to 60 pg/mL (Stage 3 subjects) or greater than or equal to 90 pg/mL (Stage 4 subjects).
  * An adjusted serum calcium value greater than or equal to 8.2 mg/dL (2.05 mmol/L) to less than or equal to 10.5 mg/dL (2.63 mmol/L).
  * A serum phosphorus value greater than or equal to 2.0 mg/dL (0.65 mmol/L but less than or equal to 6.0 mg/dL (1.94 mmol/L).
* For entry into the Treatment Phase (vitamin D receptor activator naïve subjects and those that have completed a 4 week washout), the subject must have:

  * iPTH measurement that is greater than or equal to 75 pg/mL (Stage 3 subjects) or greater than or equal to 110 pg/mL (Stage 4 subjects).
  * An adjusted serum calcium value greater than or equal to 8.4 mg/dL (2.10 mmol/L) but less than or equal to 10.2 mg/dL (2.55 mmol/L).
  * A serum phosphorus value greater than or equal to 2.5 mg/dL (0.81 mmol/L) but less than or equal to 5.8 mg/dL (1.87 mmol/L).
  * Must have 25-hydroxyvitamin D levels ≥ 30 ng/mL prior to washout, if not VDRA naïve, or treatment in Part II of the study.

Exclusion Criteria:

* All subjects that have had a small bowel transplant will be excluded from the study.
* Subject has had acute kidney failure within 12 weeks of the Screening Phase (defined as an acute rise in serum creatinine).
* Subject has had symptomatic or significant hypocalcemia requiring active vitamin D therapy (for example, calcitriol, paricalcitol, doxercalciferol or alfacalcidol) within 6 months prior to the Screening Phase.
* Subject has a history of active kidney stones (6 months prior to screening).
* Subject has chronic gastrointestinal disease, which in the investigator's opinion may cause significant gastrointestinal malabsorption.
* Subject is taking maintenance calcitonin, bisphosphonates, cinacalcet, glucocorticoids in an equivalent dose of greater than 5 mg prednisone daily, or other drugs known to affect calcium or bone metabolism within 4 weeks prior to treatment.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2010-02; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Chand, MD, Study Director — AbbVie

REFERENCES:
- [Result] Webb NJA, Lerner G, Warady BA, Dell KM, Greenbaum LA, Ariceta G, Hoppe B, Linde P, Lee HJ, Eldred A, Dufek MB. Efficacy and safety of paricalcitol in children with stages 3 to 5 chronic kidney disease. Pediatr Nephrol. 2017 Jul;32(7):1221-1232. doi: 10.1007/s00467-017-3579-6. Epub 2017 Mar 22. PMID 28332096
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 was an open-label, single-dose study evaluating the pharmacokinetics of paricalcitol capsules in children with moderate to severe chronic kidney disease (CKD). Part 2 consisted of a double-blind, placebo-controlled study to evaluate safety and efficacy of paricalcitol and an open-label phase where all participants received paricalcitol.
Pre-assignment Details: Two participants enrolled in Part 2 after completing Part 1 of the study, hence the actual total number of enrolled participants is equal to 47.
Period: Part 1
Arm/Group | Part 1: Paricalcitol | Part 2: Placebo | Part 2: Paricalcitol
Started | 12 | 0 | 0
Completed | 12 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part 2 Double-blind Treatment Period
Arm/Group | Part 1: Paricalcitol | Part 2: Placebo | Part 2: Paricalcitol
Started | 0 | 18 (Includes one participant who enrolled in Part 2 after completing Part 1) | 19 (Includes one participant who enrolled in Part 2 after completing Part 1)
Received Treatment | 0 | 18 | 18
Completed | 0 | 16 | 13
Not Completed | 0 | 2 | 6
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Required a Dose Reduction | 0 | 0 | 3
Not completed — Randomized in Error | 0 | 0 | 1
Period: Part 2 Open-label Period
Arm/Group | Part 1: Paricalcitol | Part 2: Placebo | Part 2: Paricalcitol
Started | 0 | 16 | 13
Completed | 0 | 12 | 12
Not Completed | 0 | 4 | 1
Not completed — Adverse Event | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants. Note: Two participants enrolled in Part 2 after completing Part 1 of the study, hence the actual total number of enrolled participants was 47. These 2 participants are counted in both arms they enrolled in for Baseline Measure data and are hence double-counted in the Total column for gender, race and CKD stage.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Paricalcitol | Part 2: Placebo | Part 2: Paricalcitol | Total
Number analyzed (Participants) | 12 | 18 | 19 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline measure data were analyzed separately for participants in Part 1 and Part 2.
  years
    Part 1: number analyzed (Participants) | 12 | 0 | 0 | 12
    Part 1 | 13.5 (1.98) |  |  | 13.5 (1.98)
    Part 2: number analyzed (Participants) | 0 | 18 | 19 | 37
    Part 2 |  | 13.3 (1.75) | 13.9 (1.81) | 13.6 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 6 | 14
  Male | 9 | 13 | 13 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 17 | 14 | 41
  Black | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 4 | 4
  American Indian/Alaska Native | 1 | 0 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  Other | 0 | 1 | 1 | 2
Chronic Kidney Disease Stage [Count of Participants; unit: Participants] — Stage 3: estimated glomerular filtration rate (eGFR) 30 to 59 mL/min/1.73 m²; Stage 4: eGFR 15 to 29 mL/min/1.73 m², not requiring dialysis
  Participants
    Stage 3 | 6 | 11 | 10 | 27
    Stage 4 | 6 | 7 | 8 | 21
    Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Paricalcitol Maximum Observed Plasma Concentration (Cmax)
Time Frame: Blood samples were collected at hour 0, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours after dosing.
Population: All participants enrolled and administered paricalcitol for the pharmacokinetic (PK) period, Part 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Paricalcitol
Number analyzed (Participants) | 12
ng/mL | 0.13 (0.052)

2. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-∞)
Time Frame: Blood samples were collected at hour 0, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours after dosing.
Population: All participants enrolled and administered paricalcitol for the PK Portion, Part 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 1: Paricalcitol
Number analyzed (Participants) | 12
ng*hr/mL | 2.87 (0.84)

3. Primary Outcome: Part 2: Percentage of Participants Achieving Two Consecutive Reductions at Least 30% From Baseline in iPTH
Description: The primary efficacy endpoint was the percentage of participants who achieved two consecutive ≥ 30% reductions from baseline in intact parathyroid hormone (iPTH) levels during the 12 week double-blind portion of the study regardless of CKD stage.
Time Frame: 12-week double-blind treatment period
Population: The Intent-To-Treat (ITT) Dataset, defined as the set of all randomized participants who took at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo | Part 2: Paricalcitol
Number analyzed (Participants) | 18 | 18
percentage of participants | 0 | 27.8
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Treatment effects were evaluated based on a two-sided significance level of 0.050. The primary efficacy analysis was a comparison between the paricalcitol capsules and placebo groups in the percentage of participants achieving 2 consecutive ≥ 30% reductions in iPTH from baseline regardless of CKD stage conducted using Fisher's exact test; Test type: Superiority or Other; p = 0.045, Fisher Exact; Difference = 27.8, 95% CI 2-sided [7.5 to 52.8]

4. Secondary Outcome: Part 2: Percentage of Participants Achieving a Final iPTH Within KDOQI Target Ranges
Description: The Kidney Disease Outcomes Quality Initiatives (KDOQI) Pediatric Subcommittee on Practice Guidelines for Bone Metabolism and Disease in Children with CKD target range for intact parathyroid hormone (iPTH) is as follows::
  CKD Stage 3: 35 - 69 pg/mL; CKD Stage 4: 70 - 110 pg/mL.
Time Frame: Week 12
Population: Intent to treat dataset
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo | Part 2: Paricalcitol
Number analyzed (Participants) | 18 | 18
percentage of participants | 11.1 | 33.3
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Test type: Superiority or Other; p = 0.128, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CHM) test, adjusting for CKD Stage

5. Secondary Outcome: Part 2: Change From Baseline in iPTH to Each Post-baseline Visit
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Intent to treat dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Part 2: Placebo | Part 2: Paricalcitol
Number analyzed (Participants) | 18 | 18
pg/mL
  Week 2: number analyzed (Participants) | 15 | 16
  Week 2 | 50.39 (15.186) | -12.16 (14.695)
  Week 4: number analyzed (Participants) | 18 | 16
  Week 4 | 57.16 (20.813) | -11.27 (22.117)
  Week 8: number analyzed (Participants) | 18 | 13
  Week 8 | 57.31 (22.099) | -12.79 (24.814)
  Week 12: number analyzed (Participants) | 15 | 12
  Week 12 | 71.47 (17.661) | -17.05 (19.186)
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Overall Comparison (all time points): A mixed effects repeated measures analysis using all the longitudinal observations across the visits including the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, and the continuous covariate of baseline measurement; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Differenbce = -72.40, 95% CI 2-sided [-108.05 to -36.75]
Statistical Analysis 2: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Week 2 Comparison: a mixed effects repeated measures analysis using all the longitudinal observations across the visits including the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, and the continuous covariate of baseline measurement; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Difference = -62.55, 95% CI 2-sided [-105.60 to -19.49]
Statistical Analysis 3: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Week 4 Comparison: a mixed effects repeated measures analysis using all the longitudinal observations across the visits including the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, and the continuous covariate of baseline measurement; Test type: Superiority or Other; p = 0.032, Mixed Models Analysis; Difference = -68.43, 95% CI 2-sided [-130.39 to -6.47]
Statistical Analysis 4: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Week 8 Comparison: A mixed effects repeated measures analysis using all the longitudinal observations across the visits including the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, and the continuous covariate of baseline measurement; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis; Difference = -70.09, 95% CI 2-sided [-137.82 to -2.37]
Statistical Analysis 5: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Week 12 Comparison: A mixed effects repeated measures analysis using all the longitudinal observations across the visits including the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, and the continuous covariate of baseline measurement; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Difference = -88.52, 95% CI 2-sided [-142.04 to -35.01]

6. Secondary Outcome: Part 2: Percentage of Participants Achieving Final Calcium Levels Within KDOQI Target Ranges
Description: KDOQI recommends serum calcium is maintained within age appropriate normal ranges:
  Age 6 - 12: 9.4 - 10.2 mg/dL (2.35 - 2.55 mmol/L); Age 13 - 20: 8.8 - 10.2 mg/dL (2.20 - 2.55 mmol/L).
Time Frame: Week 12
Population: Intent to treat dataset
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo | Part 2: Paricalcitol
Number analyzed (Participants) | 18 | 18
percentage of participants | 94.4 | 83.3
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Test type: Superiority or Other; p = 0.327, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CHM) test, adjusting for CKD Stage

7. Secondary Outcome: Part 2: Percentage of Participants Achieving Final Phosphorus Levels Within KDOQI Target Ranges
Description: The KDOQI target ranges of serum phosphorus are to maintain at or above age appropriate lower limits and no higher than the age-appropriate upper limits:
  Age 6 - 12: 3.6 - 5.8 mg/dL (1.16 - 1.87 mmol/L); Age 13 - 20: 2.3 - 4.5 mg/dL (0.74 - 1.45 mmol/L).
Time Frame: Week 12
Population: Intent to treat dataset
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo | Part 2: Paricalcitol
Number analyzed (Participants) | 18 | 18
percentage of participants | 72.2 | 50.0
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; Test type: Superiority or Other; p = 0.194, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CHM) test, adjusting for CKD Stage

8. Secondary Outcome: Part 2: Change From Baseline in First Morning Void (FMV) Urinary Albumin to Creatinine Ratio (UACR)
Description: The mean change from Baseline in FMV UACR on a log scale to each post baseline visit.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: Intent-to-treat dataset with available Baseline data, and available data at each time point
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | Part 2: Placebo | Part 2: Paricalcitol
Number analyzed (Participants) | 15 | 16
mg/g
  Week 4: number analyzed (Participants) | 15 | 13
  Week 4 | -0.12 (0.126) | -0.13 (0.132)
  Week 8: number analyzed (Participants) | 14 | 11
  Week 8 | -0.13 (0.141) | -0.01 (0.155)
  Week 12: number analyzed (Participants) | 12 | 10
  Week 12 | -0.08 (0.259) | 0.22 (0.292)
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.469, Mixed Models Analysis; Difference = 0.14, 95% CI 2-sided [-0.25 to 0.53]
Statistical Analysis 2: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.975, Mixed Models Analysis; Difference = -0.01, 95% CI 2-sided [-0.39 to 0.37]
Statistical Analysis 3: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p = 0.567, Mixed Models Analysis; Difference = 0.12, 95% CI 2-sided [-0.32 to 0.56]
Statistical Analysis 4: Comparison: Part 2: Placebo vs Part 2: Paricalcitol; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.462, Mixed Models Analysis; Difference = 0.30, 95% CI 2-sided [-0.53 to 1.12]

ADVERSE EVENTS:
Time Frame: Part 1: From the time of study drug administration through 30 days following the single dose of study drug. Part 2 Double-blind Period: From the first dose of study drug until the last dose of study drug during the double-blind period (12 weeks). Part 2 Open-label Period: From the first dose during the open-label period until 30 days after the last dose of study drug during the open-label period (up to 16 weeks).
Groups:
- Part 2: Placebo: Participants received placebo capsules three times a week for 12 weeks during the double-blind treatment phase.
- Part 2: Paricalcitol: Participants received paricalcitol three times a week (TIW) for 12 weeks during the double-blind treatment period. The initial dose of paricalcitol was 1 µg TIW. Doses could be adjusted based on chemistry evaluations to target Kidney Disease Outcomes Quality Initiatives (KDOQI) levels.
- Part 2: Placebo/Paricalcitol: Participants who received placebo in the double-blind treatment phase received open-label paricalcitol at an initial dose of 1 µg three times a week in the open- label treatment phase (Weeks 12-24). Doses could be adjusted based on chemistry evaluations to target KDOQI levels.
- Part 2: Paricalcitol/Paricalcitol: Participants who received paricalcitol during the double-blind treatment period continued to receive paricalcitol three times a week during the open-label period (Weeks 12-24).
Arm/Group | Part 1: Paricalcitol | Part 2: Placebo | Part 2: Paricalcitol | Part 2: Placebo/Paricalcitol | Part 2: Paricalcitol/Paricalcitol
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/18 | 0/18 | 1/16 | 1/13
Other Adverse Events (participants affected / at risk) | 2/12 | 15/18 | 7/18 | 12/16 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Paricalcitol (N=12) | Part 2: Placebo (N=18) | Part 2: Paricalcitol (N=18) | Part 2: Placebo/Paricalcitol (N=16) | Part 2: Paricalcitol/Paricalcitol (N=13)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
HOMICIDAL IDEATION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Paricalcitol (N=12) | Part 2: Placebo (N=18) | Part 2: Paricalcitol (N=18) | Part 2: Placebo/Paricalcitol (N=16) | Part 2: Paricalcitol/Paricalcitol (N=13)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
FEELING HOT (General disorders) | 0 | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 1 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 0 | 1 | 0
IMPETIGO (Infections and infestations) | 0 | 0 | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 2 | 0 | 1 | 2
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PARONYCHIA (Infections and infestations) | 0 | 1 | 0 | 0 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 2 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 3 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 2 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 2 | 0 | 0 | 0
INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
VITAMIN D DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 0
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 1 | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
THINKING ABNORMAL (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.